CLINICAL TRIAL: NCT01102088
Title: Phase I/II Study of Evaluating the Safety and Efficacy of Using a Simultaneous Integrated Boost for Dose Escalation in Patients With Esophageal Cancer
Brief Title: Simultaneous Integrated Boost (SIB) in Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0847; NCI-2011-02030 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-04-09; First posted 2010-04-12 (Estimated); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Esophageal Cancer
Keywords: Cancer; Gastroesophageal; Simultaneous Integrated Boost; SIB; 5-Fluorouracil; 5-FU; Adrucil; Efudex; Docetaxel; Taxotere; Radiation; chemoradiation
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation + Chemotherapy (Experimental): Simultaneous integrated boost (SIB) used in combination with a fixed dose of radiation (180 cGy in 28 fractions = 5040 Gy PTV dose). Two dose levels (210 cGy and 225 cGy each in 28 fractions) of SIB will be considered in the phase I part of the study, starting at 210 cGy in 28 daily fractions.
  For the phase II part of the study once the MTD has been achieved proton therapy will be allowed. Treatment dose will be identical to that of the photon treatment where the PTV is treated to 50.4 Gy(RBE) (RBE=1.1) while the CTV is boosted to 63 Gy(RBE) in 28 fractions.
  Chemotherapy Administration: Schedule of chemotherapy, and modifications of chemotherapy drugs during chemoradiation treatment will be at the discretion of the treating medical oncologist per their standard of practice and with consideration to standard chemotherapy drugs in the treatment of esophageal cancer.
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Simultaneous integrated boost (SIB) used in combination with a fixed dose of radiation (180 cGy in 28 fractions = 5040 Gy PTV dose). Two dose levels (210 cGy and 225 cGy each in 28 fractions) of SIB will be considered in the phase I part of the study, starting at 210 cGy in 28 daily fractions.
  For the phase II part of the study once the MTD has been achieved proton therapy will be allowed. Treatment dose will be identical to that of the photon treatment where the PTV is treated to 50.4 Gy(RBE) (RBE=1.1) while the CTV is boosted to 63 Gy(RBE) in 28 fractions.

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of radiation that can be given in combination with chemotherapy in patients with esophageal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
Radiation Therapy:

If you are found to be eligible, you will receive radiation therapy 5 days for 5 weeks. On Week 6, you will receive radiation therapy on 3 days. You will be assigned to a dose level of radiation based on when you join this study. Up to 2 dose levels of radiation will be tested. The first group of participants will receive the lower dose level. The next group will receive a higher dose than the group before it, if no intolerable side effects were seen.

Chemotherapy Administration:

Your medical oncologist and or his/her team will review and discuss all aspects of chemotherapy administration including drugs you will receive, schedule of chemotherapy, and their side effects with you before starting treatment.

Your study doctor may adjust your chemotherapy dose if you experience intolerable side effects.

Study Visits:

You will have weekly study visits while you are receiving radiation therapy. You may have an extra study visit if your doctor thinks it is necessary. At each visit:

* Your complete medical history will be recorded.
* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will be asked how you are feeling and about any side effects you may be having.
* Blood ( about 2-3 teaspoons) will be drawn for routine tests.

Length of Study:

You will receive radiation and chemotherapy for up to 6 weeks. You will be taken off study if the disease gets worse or if you experience intolerable side effects.

Visit After the Last Dose:

You will have a study visit 2 weeks (+/- 5 days) after you stop receiving radiation. If you are unable to return to MD Anderson, most of this may be done over the phone. At this visit:

* Your complete medical history will be updated.
* You will be asked how you are feeling and about any side effects that you may be having.
* If the doctor feels it is necessary you will have a physical exam, including measurement of your weight, vital signs, and your performance status will be recorded. If you are unable to travel to this visit, you will not have a physical exam.

Follow-Up Visits:

Your will have follow-up visits after 4 weeks from completing your radiation treatments. Your doctor will decide when you are to return and which tests and procedures will be performed. The following tests and procedures may be performed:

* Your complete medical history may be recorded.
* You may have a physical exam, including measurement of your weight and vital signs.
* You may have a CT or PET scan to check the status of the disease.
* You may be asked how you are feeling and about any side effects you may be having.
* You may have an upper GI endoscopy with biopsies.

If the study doctor thinks it is needed, every year (+/- 2 months), the following tests and procedures will be performed to check the status of the disease:

* You will have a CT or PET/CT scan.
* You may have an upper endoscopy and tumor biopsy.

This is an investigational study. The chemotherapy agents are FDA approved and are commercially available for use in the treatment of esophageal cancer. The higher dose level of radiation in this study is considered investigational.

Up to 42 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed primary (non-recurrent) adenocarcinoma (AC) or squamous cell carcinoma of the esophagus or AC of the gastroesophageal (GE) junction.
2. Age >/= 18.
3. Patients must be deemed unresectable disease or considered for a selective surgical approach (where surgery is delay if a patient achieves a complete response) as determined by the multidisciplinary evaluation or patient is not considered operable due to medical reasons.
4. Patients with distant metastasis and life expectancy >/= 3 months are eligible.
5. ECOG Performance Status 0-2
6. No prior radiation to the thorax that would overlap with the current treatment field, prior radiation to other areas is allowed.
7. Patients with nodal involvement are eligible
8. Adequate bone marrow, and renal functions as assessed by the following: Hemoglobin >/= 9.0 g/dl, Platelet count >/= 100,000/mm^3, Creatinine </=1.5 times ULN
9. Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
10. Patients (men and women) of childbearing potential must use effective method of birth control throughout their participation in this study.
11. Induction chemotherapy is allowed.

Exclusion Criteria:

1. Patients with T1, N0 lesions.
2. Patients with a TE fistula or direct invasion into the mucosa of the trachea or major bronchi. Bronchoscopy is encouraged if a TE fistula is suspected. The presence of a fistula will exclude a patient from this study.
3. Prior surgery or radiotherapy for esophageal or gastroesophageal junction cancer.
4. Prior radiotherapy that would overlap the anticipated study treatment fields.
5. Patients with active second malignancy are allowed as long as it is determined that the treatment of esophageal cancer is a higher priority through proper subspecialty consultations.
6. Uncontrolled concurrent illness including, but not limited to: serious uncontrolled infection, symptomatic congestive heart failure (CHF), unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with the study requirements.
7. Known hypersensitivity to docetaxel, 5-FU.
8. Any other condition or circumstance that would, in the opinion of the Investigator, make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2019-06-08 (Actual); Study Completion 2019-06-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Simultaneous Integrated Boost (SIB) | 8 Weeks
  MDT defined as CTCAE 3 grade 3 acute radiation toxicity of esophagitis 2 weeks after completion of 6 weeks of radiation therapy.

SECONDARY OUTCOMES:
Time to Local Failure | 1 year
  Local control assessed radiographically using either a PET or CT scan. The one-year local failure rate monitored using the methods of Thall et al.
Pathologic Response | 2 months after radiation therapy
  Complete pathologic response defined as no gross or microscopic tumor in the surgical specimen using light microscopy, but not immunohistochemical stains. Tissue from esophagogastroduodenoscopy can also be used. A partial pathologic response defined as shrinkage in tumor size compared with the original esophagogastroduodenoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: James Welsh, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chen D, Menon H, Verma V, Seyedin SN, Ajani JA, Hofstetter WL, Nguyen QN, Chang JY, Gomez DR, Amini A, Swisher SG, Blum MA, Younes AI, Barsoumian HB, Erasmus JJ, Lee JH, Bhutani MS, Hess KR, Minsky BD, Welsh JW. Results of a Phase 1/2 Trial of Chemoradiotherapy With Simultaneous Integrated Boost of Radiotherapy Dose in Unresectable Locally Advanced Esophageal Cancer. JAMA Oncol. 2019 Nov 1;5(11):1597-1604. doi: 10.1001/jamaoncol.2019.2809. PMID 31529018
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org